CLINICAL TRIAL: NCT03596255
Title: Clinical Estimation of Dental Anxiety
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Markus Höglund, PHD-student, specialist in orofacial medicin, Doctor of Dental Surgery, Karolinska Institutet
Other Study IDs: 0001
Record Dates: First submitted 2018-06-27; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: All public dental clinics in the region of Östergötland, Sweden, were asked to consecutively recruit adult patients returning for their annual examination
  Interventions: Diagnostic Test: MDAS
- Dental personnel: All public dental clinics in the region of Östergötland, Sweden were contacted and asked to participate in the study
  Interventions: Diagnostic Test: Estimated level of DA

INTERVENTIONS:
Diagnostic Test: Estimated level of DA — the dental personnel estimated the patient's level of DA (eDA) on a 100mm VAS
  Groups: Dental personnel
Diagnostic Test: MDAS — The patient rated their DA using the Modified Dental Anxiety Scale (MDAS)
  Groups: Patients

SUMMARY:
Introduction: Dental anxiety (DA) is treatable and preventable when dental personnel correctly estimate the patient's level of DA. Objective: To evaluate dental personnel's ability to estimate DA.

DETAILED DESCRIPTION:
Method: All public dental clinics in the region of Östergötland, Sweden, were asked to consecutively recruit adult patients returning for their annual examination. The patient rated DA using the Modified Dental Anxiety Scale (MDAS) and a Visual Analogue Scale of dental anxiety (DA-VAS). The patient also recorded gender, age, level of education and confidence in handling DA. After the examination, the dental personnel estimated the patient's level of DA (eDA) on a VAS. The examiner also recorded gender, age, profession, years of experience, country of education, interest in DA, special education concerning DA and confidence in ability to handle DA.

ELIGIBILITY:
Inclusion Criteria:

Adult patients returning for their annual examination on a public dental clinics in the region of Östergötland, Sweden during a two week period.

Exclusion Criteria:

inability to fill in the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients returning for their annual examination on a public dental clinics in the region of Östergötland, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Estimated Dental anxiety on a 100mm VAS vs MDAS | through study completion, 2 weeks/clinic and a total of aproximatly 6 months
  The dental personnel's Clinical estimation of how dentally anxious their patient are (where 0mm represent minimal and 100mm maximal.) compared to the patients one rating of dental anxiety(Measured whit the Modified Dental Anxiety Scale(MDAS) where 5 is minimal and 25 maximal) .

SECONDARY OUTCOMES:
The patients Dental Anxiety, measured whit the "Modified Dental Anxiety Scale"(MDAS) | through study completion, 2 weeks/clinic and a total of approximately 6 months
  The Patients own ration of how dentally anxious they are. Measured whit the Modified Dental Anxiety Scale(MDAS) where 5 is minimal and 25 maximal

CONTACTS AND LOCATIONS:
Overall Officials: Mats Bågesund, Lecturer, Study Director — Linköpings University, Sweden.
Locations (1):
- Centrum för Orofacial Medicin, Torkelbergsgatan 11., Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will only be presented at group level.